CLINICAL TRIAL: NCT06520709
Title: Kinesiophobia and Associated Factors in Postmenopausal Osteoporosis: A Controlled Study
Brief Title: Kinesiophobia in Postmenopausal Osteoporosis
Status: Completed | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, MD, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH1
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Osteoporosis
Keywords: osteoporosis; quality of life; kinesiophobia; depression; anxiety
MeSH Terms: conditions — Osteoporosis; Kinesiophobia; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postmenopausal osteoporosis: Postmenopausal osteoporosis
  Interventions: Other: No intervention
- Control group: Healthy group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aims to evaluate kinesiophobia levels in postmenopausal women with osteoporosis compared to a healthy control group and to explore the relationships between kinesiophobia and various psychosocial factors, including quality of life, fear of falling, and symptoms of depression and anxiety.

DETAILED DESCRIPTION:
This cross-sectional, controlled study aims to explore kinesiophobia levels in postmenopausal women with osteoporosis compared to healthy age-matched controls. Postmenopausal osteoporosis is a systemic condition characterized by reduced bone mineral density, which increases fracture risk and can significantly affect individuals' physical activity and overall quality of life. Kinesiophobia, or the irrational fear of movement due to perceived injury risk, can further exacerbate this issue by restricting physical activity, which is vital for maintaining bone health. The study will involve 60 postmenopausal women diagnosed with osteoporosis and 60 healthy age-matched women without osteoporosis or osteopenia. Participants will be recruited from the outpatient clinics of İstanbul Physical Therapy and Rehabilitation Training and Research Hospital between January 21, 2024, and February 21, 2024. The study will assess kinesiophobia using the Turkish version of the Tampa Scale for Kinesiophobia (TSK), quality of life with the Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41), and symptoms of depression and anxiety using the Hospital Anxiety and Depression Scale (HADS). Additionally, the Tinetti Falls Efficacy Scale (TFES) will evaluate fear of falling, and bone mineral density will be measured using dual-energy X-ray absorptiometry (DXA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Participants must be diagnosed with postmenopausal osteoporosis and have been under follow-up for at least six months.
* Age: Individuals must be 50 years or older.
* Health Status: Participants must have excluded secondary causes of osteoporosis.

Exclusion Criteria:

* Comorbid Conditions: Presence of other musculoskeletal, neurological, or psychiatric diseases that could influence kinesiophobia or pain.
* Cognitive or Communication Difficulties: Any cognitive dysfunction or communication issues that might impair the participant's ability to engage with the study.
* Acute Conditions: Presence of acute painful conditions that might affect the results.
* Medications: Use of medications or presence of diseases that could cause balance or functional disorders.

Min Age: 50 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Osteoporosis Group: This group included 60 postmenopausal women diagnosed with osteoporosis. Participants were required to have been under follow-up for at least six months.
  Control Group: This group comprised 60 healthy postmenopausal women who were neither osteoporotic nor osteopenic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK) | 0 day
  The Tampa Scale for Kinesiophobia (TSK) is a widely used tool for assessing fear of movement and physical activity, often referred to as kinesiophobia.

SECONDARY OUTCOMES:
Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41) | 0 day
  The Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41) is a comprehensive instrument specifically designed to assess the quality of life in individuals with osteoporosis
Hospital Anxiety and Depression Scale (HADS) | 0 day
  The Hospital Anxiety and Depression Scale (HADS) is a widely used tool for assessing levels of anxiety and depression in patients, particularly in medical settings.
Tinetti Falls Efficacy Scale (TFES) | 0 day
  The Tinetti Falls Efficacy Scale (TFES) is a tool designed to assess an individual's fear of falling and their perceived confidence in their ability to perform various activities without falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No